CLINICAL TRIAL: NCT04681638
Title: Plasma Resuscitation withOut Lung Injury
Acronym: PROPOLIS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment targets were unable to be reached due to difficulty in locating and contacting the Legally Authorized Representative (LAR). Even with prolonged enrollment timeframe, the study was unable to obtain consent from the LAR.
Sponsor: Coalition for National Trauma Research (Other)
Collaborators: Cerus Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNTR-2020-001; CDMRP-DM190167 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2020-12-04; First posted 2020-12-23 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Burns
MeSH Terms: conditions — Burns | interventions — Crystalloid Solutions

STUDY DESIGN:
Intervention Model Description: This is an open-label, phase IV, multicenter, randomized controlled prospective clinical trial in patients with burns. The study model is parallel (between-patient). The intervention to be tested is Pathogen-Reduced Plasma for burn shock resuscitation vs. standard-of-care resuscitation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Plasma (Experimental): Pathogen-Reduced Plasma resuscitation
  Interventions: Drug: Pathogen-Reduced Plasma
- Crystalloid (Active Comparator): Standardized crystalloid resuscitation
  Interventions: Drug: Crystalloid Solutions

INTERVENTIONS:
Drug: Pathogen-Reduced Plasma — The treatment group will receive an additional infusion of Pathogen-Reduced Plasma based on the formula, hourly rate, mL/hr = (1 mL*kg*TBSA)/24 hr. This infusion will not be titrated. It will be discontinued at the end of the 24th postburn hour.
  Other Names: PRP
  Arms: Plasma
Drug: Crystalloid Solutions — The control group will receive an additional infusion of LR based on the formula: hourly rate, mL/hr = (1mL*kg*TBSA)/24 hr. this infusion will not be titrated. It will be discontinued at the end of the 24th postburn hour.
  Other Names: LR
  Arms: Crystalloid

SUMMARY:
The treatment of patients with major burns requires resuscitation with massive amounts of fluid, typically a type of salt water that is given by vein. This frequently results in injury to vital organs, especially the lungs and kidneys, and even in death. In this study, the investigators propose to use plasma, a specially prepared blood product made from the liquid part of blood, that has undergone special treatment to reduce the risk of disease transmission. The aims include 1) reduce the amount of fluid given during the first 24 hours after a burn 2) reduce the incidence of lung injury and other complications related to the administration of funds and 3) determine if the blood product has any effect on inflammation. An overall decrease the amount of fluids that burn patients receive should decrease the potential for lung injury, decrease days in the hospital, and improve survival.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Weight > 40 kg
* Initial assessment of thermal injury size ≥ 20% TBSA
* Admitted to the burn center and enroll able within 8 hours of injury
* Expected to receive intravenous resuscitation fluids for at least 24 hours after injury
* Expected to live > 24 hours after injury

Exclusion Criteria:

* Chemical injury
* Deep electric injury
* Associated non-thermal injuries with estimated Injury Severity Score > 25
* Inability to obtain informed consent
* Decision not to treat due to injury severity or other factors
* Patient age > 65 years or < 18 years
* Presence of anoxic brain injury that is not expected to result in complete recover
* Patent already receiving plasma infusion, or judged to be likely to require plasma infusion
* Patent already receiving "rescue procedures" (albumin infusion, CRRT, TPE, or high-dose ascorbic acid)
* Existence of pre-morbid conditions: Congestive heart failure (NYHA Class IV); End-stage kidney disease (dialysis patient); Cirrhosis of the liver; Oxygen-dependent chronic obstructive pulmonary disease; Malignancy currently under treatment; Previous bilateral lower extremity amputations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2022-08-17 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-09-29 (Actual)

PRIMARY OUTCOMES:
The total volume of all resuscitation fluids delivered between hours 0-24 postern, in ml/kg. | 24 hours
  The total volume of all resuscitation fluids delivered between hours 0-24 postburn, in ml/kg

SECONDARY OUTCOMES:
Total resuscitation volume in ml/kg | 48 hours
  The total volume of all resuscitation fluids delivered between hours 0-48 postburn, in ml/kg
Total 24 hour resuscitation volume in ml/kg/TBSA | 24 hours
  The total volume of all resuscitation fluids delivered between hours 0-24 postburn, in ml/kg/TBSA
Total 48 hour resuscitation volume in ml/kg/TBSA | 48 hours
  The total volume of all resuscitation fluids delivered between hours 0-48 postburn, in ml/kg/TBSA
Hemodynamic instability | 48 hours
  Severity and duration of hemodynamic instability during hours 0-48 postburn (norepinephrine equivalents)
Metabolic acidosis | 48 hours
  Severity and duration of metabolic acidosis (arterial lactate levels)
Incidence of "rescue" (a) | 48 hours
  Initiation of extracorporeal therapy (continuous renal replacement therapy or therapeutic plasma exchange
Incidence of "rescue" (b) | 48 hours
  Infusion of high-dose ascorbic acid (66 mg/kg/hr)
Incidence of "rescue" (c) | 24 hours
  Initiation of a continuous infusion of albumin
Acute Respiratory Distress Syndrome | 7 days
  Incidence of Acute Respiratory Distress Syndrome using Berlin Criteria
Mechanical ventilation | 28 days
  Ventilator free days
Intensive Care Unit days | 28 days
  Intensive Care Unit free days
Multi-Organ Failure Assessment | 7 days
  Sequential Organ Failure Assessment scores. Minimum score 1, maximum score 4. The higher the score the worse the outcome.
Transfusion-Related Acute Lung Injury | 72 hours
  Incidence of Transfusion-Related Acute Lung Injury, Type I or II.
Thromboembolic events | 7 days
  Incidence of venous thrombosis-embolic events (deep vein thrombosis or pulmonary embolism)
Mortality | throughout study completion, an average of 1 year
  In hospital mortality
Patient reported outcomes | 6 months
  Patient reported outcomes using the Patient Reported Outcomes Measurement Information System, Global 10. This scale10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. Higher scores equal a healthier patient.
Syndecan-1 levels | 48 hours
  Syndecan-1 level in ng/dl
Cytokines | 48 hours
  Cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Leopoldo Cancio, MD, Principal Investigator — U.S. Army Burn Center
Locations (6):
- United States (6):
  - University of Alabama at Birmingham Burn Center, Birmingham, Alabama
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - U.S. Army Burn Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Washington School of Medicine, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available one year after initial results publication.